CLINICAL TRIAL: NCT06651229
Title: A Phase 1, First-in-Human, Dose Escalation Study of JNJ-90189892 for Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Neoplasms
Brief Title: A Study of JNJ-90189892 for Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 90189892AML1001; 90189892AML1001 (Other: Janssen Research & Development, LLC); 2024-514341-10-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Neoplasms
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-90189892 (Experimental): Participants will receive JNJ-90189892 in Part 1 (Dose escalation) of the study and the dose levels will be escalated sequentially based on the decisions of the study evaluation team (SET) until the recommended phase 2 dose (RP2D) has been identified. Participants in Part 2 (Dose expansion) will receive JNJ-90189892 at the RP2D determined in Part 1.
  Interventions: Drug: JNJ-90189892

INTERVENTIONS:
Drug: JNJ-90189892 — JNJ-90189892 will be administered.

SUMMARY:
The purpose of Part 1 (Dose Escalation) of the study is to assess the effective dose (recommended Phase 2 dose[s] [RP2Ds]) that can be safely administered, and dosing regimens of JNJ-90189892 in participants with relapsed or refractory (R/R) acute myeloid leukemia (AML) or R/R higher-risk type of myelodysplastic neoplasms (type of cancer of the blood and bone marrow, which does not respond to treatment or comes back after treatment). The purpose of Part 2 (Cohort Expansion) is to further assess the safety, tolerability and efficacy in participants with R/R AML or higher-risk types of MDS.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis, per the world health organization (WHO) 2022 criteria, of (a) Acute myeloid leukemia (AML) or (b) Moderate high, high, or very high-risk myelodysplastic neoplasms (MDS) per Molecular International Prognostic Scoring System (IPSS-M)
* Body weight that is greater than or equals to (>=) 40 kg
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Have adequate renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Estimated Glomerular Filtration Rate (eGFR) >=40 milligrams per minute (mL/min) computed with the calculator on the CKD-EPI website
* Participants must have laboratory parameters in the required range

Exclusion Criteria:

* Has a medical history of clinically significant pulmonary compromise, particularly the current need for supplemental oxygen use to maintain adequate oxygenation
* Has evidence of uncontrolled systemic viral, bacterial, or fungal infection. Antimicrobial prophylaxis is permitted
* Has known allergies, hypersensitivity, or intolerance to JNJ-90189892 or its excipients
* Had major surgery or had significant traumatic injury within 14 days of planned first dose of JNJ-90189892
* Had a prior or concurrent second malignancy with natural history or treatment likely to interfere with any study endpoints of safety or the efficacy of the study treatment
* Has known active central nervous system involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-08-05 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AEs) by Severity | From screening untill 30 days after last dose of study drug (that is approximately 2.5 years)
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLTs) | At least 14 days
  DLT is defined as any toxicity that requires discontinuation of treatment, any Grade 5 toxicity; Non-hematologic toxicity (Grade 3 or 4) and Hematologic toxicity.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-90189892 | Up to approximately 2.5 years
  Serum samples will be analyzed to determine concentrations of JNJ-90189892.
Area Under the Curve Over a Dosing Interval (AUC tau) of JNJ-90189892 | Up to approximately 2.5 years
  AUC tau is the total observed plasma concentration of JNJ-90189892 in the body during the time between doses. AUCtau of JNJ-90189892 will be reported.
Maximum Observed Plasma Concentration (Cmax) of JNJ-90189892 | Up to approximately 2.5 years
  Cmax is the maximum observed plasma concentration of JNJ-90189892. Cmax of JNJ-90189892 will be reported.
Minimum Observed Plasma Concentration (Cmin) of JNJ-90189892 | Up to approximately 2.5 years
  Cmin is the minimum observed plasma concentration of JNJ-90189892. Cmin of JNJ-90189892 will be reported.
Number of Participants with Presence of Anti-JNJ-90189892 Antibodies | Up to approximately 2.5 years
  Participants with presence of anti-JNJ-90189892 antibodies will be reported.
Complete Response (CR) in Acute Myeloid Leukemia (AML) | Up to approximately 2.5 years
  CR is achieved when a participant has a best response of CR (including complete response with partial hematologic recovery [CRh] or complete response with incomplete hematologic recovery [CRi]) according to the European Leukemia Network (ENL) 2022 criteria.
Overall Response (OR) in Myelodysplastic Neoplasms (MDS) | Up to approximately 2.5 years
  OR is achieved when a participant with MDS has a CR (any type, that is CRh or complete response with limited count recovery [CRL]), partial response (PR), or hematologic improvement (HI) according to the International Working Group (IWG) 2023 criteria.
Complete Response in MDS | Up to approximately 2.5 years
  CR is achieved when a participant has a best response of CR (including CRh/CRL) according to the IWG 2023 criteria.
Duration of Response (DOR) | Up to approximately 2.5 years
  DOR is defined for responsders only, as time from date of initial documentation of a response to the first documented evidence of no reponse, disease progression, relapse, initation of a new systemic anti-cancer therapy (besides hematopoietic stem cell transplant [HSCT]), or death, whichever comes first.
Time to Response (TTR) | Up to approximately 2.5 years
  TTR is defined for responders, as the time from the first dose of study drug to first qualifying response.
Number of Participants Achieving Transfusion Independence | Up to approximately 2.5 years
  Transfusion independence is defined as the absence of red blood cell (RBC) and platelet transfusions for 8 weeks or longer after starting study treatment for participants with AML and 16 weeks or longer for participants with MDS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- Australia (3):
  - Concord Hospital, Concord
  - Peter MacCallum Cancer Centre, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
- France (2):
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - Institut Claudius Regaud, Toulouse
- Spain (3):
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hospital Universitario Virgen Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency